CLINICAL TRIAL: NCT00467363
Title: The Effects of Aspirin in Gestation and Reproduction: A Multi-center, Controlled, Double-blind Randomized Trial.
Brief Title: The Effects of Aspirin in Gestation and Reproduction
Acronym: EAGeR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Enrique Schisterman, Chief and Senior Investigator, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EAGeR
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Birth; Spontaneous Abortion
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Aspirin; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): 81mg of low-dose aspirin plus 400micrograms of folic acid.
  Interventions: Drug: acetylsalicylic-acid (aspirin)
- Placebo (Placebo Comparator): 400micrograms of folic acid.
  Interventions: Dietary Supplement: Folic acid

INTERVENTIONS:
Drug: acetylsalicylic-acid (aspirin) — 81mg of low-dose aspirin plus 400micrograms of folic acid.
  Other Names: aspirin
  Arms: Aspirin
Dietary Supplement: Folic acid — 400micrograms of folic acid.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to help elucidate the effects of low-dose aspirin in combination with folic acid on the incidence of live births and spontaneous abortions among a group of women who become pregnant compared to a control group.

DETAILED DESCRIPTION:
Despite the fundamental nature of reproduction, for many it is a process fraught with frustration, inefficiency and imperfections, the effects of which can be severe. Infertility affects 10-15% of couples attempting to conceive. Among all women who conceive, the incidence of spontaneous abortion (SA) has been estimated to be between 15 and 31%, and in many cases the cause is unknown. Additionally, of the four million births yearly in the United States, between 8 and 15% will be born prematurely and experience increased morbidity and mortality as a result. An intervention with even a small absolute effect on any of these outcomes has great implications at the population level due to the large potential attributable benefit.

One such potential intervention is low-dose acetylsalicylic-acid (aspirin). Aspirin has been a primary target of interest because of its anti-inflammatory, vasodilatory and platelet aggregation inhibition properties. To evaluate the effects of low-dose aspirin in combination with folic acid on the incidence of live births and spontaneous abortion, we are conducting a multi-site randomized controlled trial study with two sites and one data coordinating center. Women aged 18-40 currently trying to become pregnant and who have had a single spontaneous abortion in the past year will be eligible for the study. The recruitment goal is 1600 women. Participating women will be randomly assigned to one of two treatment groups. Those randomized to treatment will receive daily low-dose aspirin. Those randomized to placebo will receive daily placebo. Both groups will receive folic acid daily in accordance with recommendations from the U.S. Public Health Service for prevention of birth defects. The duration of treatment regimens (LDA and folic acid or placebo and folic acid) will be 6 menstrual cycles, with those who become pregnant continuing until the end of pregnancy. Monthly urine and blood samples will be collected and questionnaires administered.

ELIGIBILITY:
Inclusion Criteria:

* Women experiencing one or two pregnancy losses at any point in gestation in the past that were not elective termination(s). At least one of these losses must be well documented by one of the following:

  * Sonogram demonstrating anembryonic loss, embryonic loss or fetal death.
  * Histologic confirmation of products of conception that were spontaneously passed per vagina or surgically obtained.
  * Hospital records of fetus delivery.
  * Late menses and positive serum hCG or positive urine hCG documented by hospital or clinic records followed by either a negative hospital/clinic pregnancy test or a decline in urinary hCG level over 3 days.
  * Home pregnancy tests without hCG confirmation from a healthcare provider (either serum or urine) will not be accepted.
* No more than 5 pregnancies in total including the pregnancy loss(es).*
* Up to two prior pregnancies that did not end in a loss.*

  *Women may have up to two pregnancies beyond 20 weeks that were not losses, two spontaneous pregnancy losses at any time in the past, and up to one therapeutic or elective termination (two therapeutic or elective terminations if no other pregnancies). Ectopic and molar pregnancies would, for the purpose of enrollment, be considered in the same category as therapeutic termination pregnancies. Women with more than two live births or those with more than two losses, regardless of the week of gestation of the loss, are excluded.
* Presence of intact tubes (both), ovaries (both), and uterus.
* Between 18 and 40 years of age at time of baseline visit.
* Regular menstrual periods between 21 - 42 days in length (within the last 12 months). Regular menstrual periods are defined as no more than an 8-day difference between the woman's shortest and longest cycle.
* No more than one missed menses in the past 12 months (other than those missed due to pregnancy or breastfeeding).
* Actively trying to conceive with a male partner and not using contraception by the baseline visit.
* Not currently pregnant at the baseline or randomization visits.
* Ability and willingness to give informed consent.
* Willingness to be randomized and to take daily study pills for 6 months to a possible 15 months

Exclusions Criteria:

* Known allergies to aspirin or non-steroidal anti-inflammatory agents.
* Clinical indication for anticoagulant therapy. These include prior or current thrombosis, antiphospholipid syndrome (APS) or known major thrombophilia.
* Clinical indication for chronic use of NSAIDs such as rheumatoid arthritis.
* Indication for additional folic acid supplementation, such as prior infant with neural tube defect (NTD), seizure disorder.
* Medical contraindication to aspirin therapy. These include uncontrolled asthma, nasal polyps, bleeding disorders, or history of gastrointestinal ulcer.
* Presence of major medical disorders (regardless of severity). These include diabetes, hypertension, systemic lupus erythematosus (SLE), untreated or active cancer (any cancer in remission or non-melanoma skin cancer is not included in the exclusion criteria), liver disease, renal disease, rheumatoid arthritis, cardiac disease, pulmonary disease other than mild asthma, neurologic disease requiring medical treatment, uncontrolled hypothyroidism, uncontrolled seizure disorder. Untreated vitamin B12 deficiency, severe anemia (Hct < 30%), hemophilia, gout, nasal polyps, among others.
* Currently undergoing/planned use of assisted reproductive techniques during trial (IVF; IUI; Clomid).
* History of infertility or sub-fertility. This includes any of the following:

  * No conception after ≥ 1 year of unprotected intercourse and actively trying to conceive.
  * Any prior medical treatment for infertility.
  * Prior treatment for known pelvic inflammatory disease.
  * Known male infertility or sperm abnormality (current partner).
  * Known tubal occlusion, anovulation, uterine abnormality, or endometriosis stage III or IV.
  * History of polycystic ovarian syndrome.
* Presence of unstable mental disorder. These include bipolar illness, schizophrenia, uncontrolled depression, uncontrolled anxiety disorder.
* Known current or recent alcohol abuse or illicit drug use.
* Current diagnosis of sexually transmitted infection (STI) (temporary exclusion)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1228 (Actual)
Dates: Start 2007-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique F Schisterman, PhD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Jean Wactawski-Wende, PhD, Principal Investigator — University at Buffalo; Robert Silver, MD, Principal Investigator — University of Utah; Noya Galai, PhD, Principal Investigator — University of Haifa; Janet Townsend, M.D., Principal Investigator — The Commonwealth Medical College; Anne Lynch, M.D., Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - University of Colorado, Denver School of Medicine, Department of Obstetrics and Gynecology, Denver, Colorado
  - Women's Health Research Center, Department of Social and Preventive Medicine, University at Buffalo, Buffalo, New York
  - Moses Taylor Hospital, Scranton, Pennsylvania
  - University of Utah Medical Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Lee IT, Barnhart KT, Hwang WT, Hinkle SN, Johnstone E, Mills JL, Caniglia EC, Schisterman EF, Mendola P, Ryan GL, Hotaling J, Peterson CM, Van Voorhis BJ, Mumford SL. Association between markers of female adiposity and live birth among patients undergoing fertility treatment or attempting unassisted conception. Hum Reprod. 2025 Sep 1;40(9):1671-1680. doi: 10.1093/humrep/deaf124. PMID 40605077
- [Derived] Freeman JR, Whitcomb BW, Bertone-Johnson ER, O'Brien LM, Dunietz GL, Purdue-Smithe AC, Kim K, Silver RM, Schisterman EF, Mumford SL. Preconception sleep, pregnancy loss, and adverse pregnancy outcomes among women with a history of pregnancy loss. Hum Reprod. 2025 Jul 1;40(7):1366-1376. doi: 10.1093/humrep/deaf074. PMID 40267399
- [Derived] Freeman JR, Whitcomb BW, Bertone-Johnson ER, O'Brien LM, Dunietz GL, Purdue-Smithe AC, Kim K, Silver RM, Schisterman EF, Mumford SL. Sleep characteristics in association with risk of sporadic anovulation among eumenorrheic women. Chronobiol Int. 2025 Apr;42(4):500-510. doi: 10.1080/07420528.2025.2481165. Epub 2025 Mar 31. PMID 40162646
- [Derived] Nobles CJ, Mendola P, Kim K, Pollack AZ, Mumford SL, Perkins NJ, Silver RM, Schisterman EF. Preconception Phthalate Exposure and Women's Reproductive Health: Pregnancy, Pregnancy Loss, and Underlying Mechanisms. Environ Health Perspect. 2023 Dec;131(12):127013. doi: 10.1289/EHP12287. Epub 2023 Dec 13. PMID 38088888
- [Derived] Nobles CJ, Mendola P, Mumford SL, Silver RM, Kim K, Perkins NJ, Schisterman EF. The Relationship of Preconception and Early Pregnancy Isoprostanes with Fecundability and Pregnancy Loss. Epidemiology. 2023 Sep 1;34(5):759-766. doi: 10.1097/EDE.0000000000001631. Epub 2023 Jul 31. PMID 37255247
- [Derived] Freeman JR, Whitcomb BW, Bertone-Johnson ER, Balzer LB, O'Brien LM, Dunietz GL, Purdue-Smithe AC, Kim K, Silver RM, Schisterman EF, Mumford SL. Preconception sleep duration, sleep timing, and shift work in association with fecundability and live birth among women with a history of pregnancy loss. Fertil Steril. 2023 Feb;119(2):252-263. doi: 10.1016/j.fertnstert.2022.10.026. Epub 2022 Dec 29. PMID 36586812
- [Derived] Schliep KC, Hinkle SN, Kim K, Sjaarda LA, Silver RM, Stanford JB, Purdue-Smithe A, Plowden TC, Schisterman EF, Mumford SL. Prospectively assessed perceived stress associated with early pregnancy losses among women with history of pregnancy loss. Hum Reprod. 2022 Sep 30;37(10):2264-2274. doi: 10.1093/humrep/deac172. PMID 35972454
- [Derived] Zolton JR, Sjaarda LA, Mumford SL, Holland TL, Kim K, Flannagan KS, Yisahak SF, Hinkle SN, Connell MT, White MV, Perkins NJ, Silver RM, Hill MJ, DeCherney AH, Schisterman EF. Preconception hemoglobin A1c concentration in healthy women is not associated with fecundability or pregnancy loss. F S Rep. 2022 Jan 20;3(1):39-46. doi: 10.1016/j.xfre.2022.01.002. eCollection 2022 Mar. PMID 35386497
- [Derived] Zhong Y, Brooks MM, Kennedy EH, Bodnar LM, Naimi AI. Use of Machine Learning to Estimate the Per-Protocol Effect of Low-Dose Aspirin on Pregnancy Outcomes: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e2143414. doi: 10.1001/jamanetworkopen.2021.43414. PMID 35262718
- [Derived] Purdue-Smithe AC, Kim K, Schliep KC, DeVilbiss EA, Hinkle SN, Ye A, Perkins NJ, Sjaarda LA, Silver RM, Schisterman EF, Mumford SL. Preconception caffeine metabolites, caffeinated beverage intake, and fecundability. Am J Clin Nutr. 2022 Apr 1;115(4):1227-1236. doi: 10.1093/ajcn/nqab435. PMID 35030239
- [Derived] Purdue-Smithe AC, Kim K, Andriessen VC, Pollack AZ, Sjaarda LA, Silver RM, Schisterman EF, Mumford SL. Preconception leukocyte telomere length and pregnancy outcomes among women with demonstrated fecundity. Hum Reprod. 2021 Nov 18;36(12):3122-3130. doi: 10.1093/humrep/deab201. PMID 34477845
- [Derived] Alkhalaf Z, Kim K, Kuhr DL, Radoc JG, Purdue-Smithe A, Pollack AZ, Yisahak SF, Silver RM, Thoma M, Kissell K, Perkins NJ, Sjaarda LA, Mumford SL. Markers of vitamin D metabolism and premenstrual symptoms in healthy women with regular cycles. Hum Reprod. 2021 Jun 18;36(7):1808-1820. doi: 10.1093/humrep/deab089. PMID 33864070
- [Derived] Naimi AI, Perkins NJ, Sjaarda LA, Mumford SL, Platt RW, Silver RM, Schisterman EF. The Effect of Preconception-Initiated Low-Dose Aspirin on Human Chorionic Gonadotropin-Detected Pregnancy, Pregnancy Loss, and Live Birth : Per Protocol Analysis of a Randomized Trial. Ann Intern Med. 2021 May;174(5):595-601. doi: 10.7326/M20-0469. Epub 2021 Jan 26. PMID 33493011
- [Derived] Mumford SL, Flannagan KS, Radoc JG, Sjaarda LA, Zolton JR, Metz TD, Plowden TC, Perkins NJ, DeVilbiss EA, Andriessen VC, A C PS, Kim K, Yisahak SF, Freeman JR, Alkhalaf Z, Silver RM, Schisterman EF. Cannabis use while trying to conceive: a prospective cohort study evaluating associations with fecundability, live birth and pregnancy loss. Hum Reprod. 2021 Apr 20;36(5):1405-1415. doi: 10.1093/humrep/deaa355. PMID 33421071
- [Derived] Flannagan KS, Mumford SL, Sjaarda LA, Radoc JG, Perkins NJ, Andriessen VC, Zolton JR, Silver RM, Schisterman EF. Is opioid use safe in women trying to conceive? Epidemiology. 2020 Nov;31(6):844-851. doi: 10.1097/EDE.0000000000001247. PMID 33311959
- [Derived] Sjaarda LA, Radoc JG, Flannagan KS, Mumford SL, Kim K, Perkins NJ, Silver RM, Schisterman EF. Urinary selective serotonin reuptake inhibitors across critical windows of pregnancy establishment: a prospective cohort study of fecundability and pregnancy loss. Fertil Steril. 2020 Dec;114(6):1278-1287. doi: 10.1016/j.fertnstert.2020.06.037. Epub 2020 Oct 14. PMID 33066974
- [Derived] Evans MB, Nobles CJ, Kim K, Hill MJ, DeCherney AH, Silver RM, Mumford SL, Sjaarda LA, Perkins NJ, Schisterman EF. Low-dose aspirin in reproductive health: effects on menstrual cycle characteristics. Fertil Steril. 2020 Dec;114(6):1263-1270. doi: 10.1016/j.fertnstert.2020.06.022. Epub 2020 Sep 4. PMID 32896390
- [Derived] Nobles CJ, Mendola P, Mumford SL, Silver RM, Kim K, Andriessen VC, Connell M, Sjaarda L, Perkins NJ, Schisterman EF. Preconception Blood Pressure and Its Change Into Early Pregnancy: Early Risk Factors for Preeclampsia and Gestational Hypertension. Hypertension. 2020 Sep;76(3):922-929. doi: 10.1161/HYPERTENSIONAHA.120.14875. Epub 2020 Aug 3. PMID 32755413
- [Derived] Hamulyak EN, Scheres LJ, Marijnen MC, Goddijn M, Middeldorp S. Aspirin or heparin or both for improving pregnancy outcomes in women with persistent antiphospholipid antibodies and recurrent pregnancy loss. Cochrane Database Syst Rev. 2020 May 2;5(5):CD012852. doi: 10.1002/14651858.CD012852.pub2. PMID 32358837
- [Derived] Yeung EH, Guan W, Zeng X, Salas LA, Mumford SL, de Prado Bert P, van Meel ER, Malmberg A, Sunyer J, Duijts L, Felix JF, Czamara D, Hamalainen E, Binder EB, Raikkonen K, Lahti J, London SJ, Silver RM, Schisterman EF. Cord blood DNA methylation reflects cord blood C-reactive protein levels but not maternal levels: a longitudinal study and meta-analysis. Clin Epigenetics. 2020 Apr 30;12(1):60. doi: 10.1186/s13148-020-00852-2. PMID 32354366
- [Derived] Russo LM, Whitcomb BW, Freeman JR, Mumford SL, Sjaarda LA, Perkins NJ, Schliep KC, Grewal J, Silver RM, Schisterman EF. Physical activity and incidence of subclinical and clinical pregnancy loss: a secondary analysis in the effects of aspirin in gestation and reproduction randomized trial. Fertil Steril. 2020 Mar;113(3):601-608.e1. doi: 10.1016/j.fertnstert.2019.10.027. PMID 32192592
- [Derived] Robinson SL, Mumford SL, Guan W, Zeng X, Kim K, Radoc JG, Trinh MH, Flannagan K, Schisterman EF, Yeung E. Maternal fatty acid concentrations and newborn DNA methylation. Am J Clin Nutr. 2020 Mar 1;111(3):613-621. doi: 10.1093/ajcn/nqz311. PMID 31858113
- [Derived] Agrawala S, Sjaarda LA, Omosigho UR, Perkins NJ, Silver RM, Mumford SL, Connell MT, Naimi AI, Halvorson LM, Schisterman EF. Effect of preconception low dose aspirin on pregnancy and live birth according to socioeconomic status: A secondary analysis of a randomized clinical trial. PLoS One. 2019 Apr 18;14(4):e0200533. doi: 10.1371/journal.pone.0200533. eCollection 2019. PMID 30998747
- [Derived] Mumford SL, Browne RW, Kim K, Nichols C, Wilcox B, Silver RM, Connell MT, Holland TL, Kuhr DL, Omosigho UR, Perkins NJ, Radin R, Sjaarda LA, Schisterman EF. Preconception Plasma Phospholipid Fatty Acids and Fecundability. J Clin Endocrinol Metab. 2018 Dec 1;103(12):4501-4510. doi: 10.1210/jc.2018-00448. PMID 30124893
- [Derived] Mumford SL, Garbose RA, Kim K, Kissell K, Kuhr DL, Omosigho UR, Perkins NJ, Galai N, Silver RM, Sjaarda LA, Plowden TC, Schisterman EF. Association of preconception serum 25-hydroxyvitamin D concentrations with livebirth and pregnancy loss: a prospective cohort study. Lancet Diabetes Endocrinol. 2018 Sep;6(9):725-732. doi: 10.1016/S2213-8587(18)30153-0. Epub 2018 May 31. PMID 29859909
- [Derived] Gibbins KJ, Mumford SL, Sjaarda LA, Branch DW, Perkins NJ, Ye A, Schisterman EF, Silver RM. Preconception antiphospholipid antibodies and risk of subsequent early pregnancy loss. Lupus. 2018 Aug;27(9):1437-1445. doi: 10.1177/0961203318776089. Epub 2018 May 17. PMID 29771194
- [Derived] Russo LM, Whitcomb BW, Mumford SL, Hawkins M, Radin RG, Schliep KC, Silver RM, Perkins NJ, Kim K, Omosigho UR, Kuhr DL, Holland TL, Sjaarda LA, Schisterman EF. A prospective study of physical activity and fecundability in women with a history of pregnancy loss. Hum Reprod. 2018 Jul 1;33(7):1291-1298. doi: 10.1093/humrep/dey086. PMID 29648647
- [Derived] Nobles CJ, Mendola P, Mumford SL, Naimi AI, Yeung EH, Kim K, Park H, Wilcox B, Silver RM, Perkins NJ, Sjaarda L, Schisterman EF. Preconception Blood Pressure Levels and Reproductive Outcomes in a Prospective Cohort of Women Attempting Pregnancy. Hypertension. 2018 May;71(5):904-910. doi: 10.1161/HYPERTENSIONAHA.117.10705. Epub 2018 Apr 2. PMID 29610265
- [Derived] Kuhr DL, Sjaarda LA, Alkhalaf Z, Omosigho UR, Connell MT, Silver RM, Kim K, Perkins NJ, Holland TL, Plowden TC, Schisterman EF, Mumford SL. Vitamin D is associated with bioavailability of androgens in eumenorrheic women with prior pregnancy loss. Am J Obstet Gynecol. 2018 Jun;218(6):608.e1-608.e6. doi: 10.1016/j.ajog.2018.03.012. Epub 2018 Mar 13. PMID 29548752
- [Derived] Sjaarda LA, Mumford SL, Kuhr DL, Holland TL, Silver RM, Plowden TC, Perkins NJ, Schisterman EF. Association of testosterone and antimullerian hormone with time to pregnancy and pregnancy loss in fecund women attempting pregnancy. Fertil Steril. 2018 Mar;109(3):540-548.e1. doi: 10.1016/j.fertnstert.2017.11.014. Epub 2018 Feb 7. PMID 29428315
- [Derived] Radin RG, Sjaarda LA, Silver RM, Nobles CJ, Mumford SL, Perkins NJ, Wilcox BD, Pollack AZ, Schliep KC, Plowden TC, Schisterman EF. C-Reactive protein in relation to fecundability and anovulation among eumenorrheic women. Fertil Steril. 2018 Feb;109(2):232-239.e1. doi: 10.1016/j.fertnstert.2017.10.025. Epub 2018 Jan 6. PMID 29317123
- [Derived] Plowden TC, Schisterman EF, Sjaarda LA, Perkins NJ, Silver R, Radin R, Kim K, Galai N, DeCherney AH, Mumford SL. Thyroid-stimulating hormone, anti-thyroid antibodies, and pregnancy outcomes. Am J Obstet Gynecol. 2017 Dec;217(6):697.e1-697.e7. doi: 10.1016/j.ajog.2017.09.001. Epub 2017 Sep 14. PMID 28917612
- [Derived] Pugh SJ, Schisterman EF, Browne RW, Lynch AM, Mumford SL, Perkins NJ, Silver R, Sjaarda L, Stanford JB, Wactawski-Wende J, Wilcox B, Grantz KL. Preconception maternal lipoprotein levels in relation to fecundability. Hum Reprod. 2017 May 1;32(5):1055-1063. doi: 10.1093/humrep/dex052. PMID 28333301
- [Derived] Sjaarda LA, Radin RG, Silver RM, Mitchell E, Mumford SL, Wilcox B, Galai N, Perkins NJ, Wactawski-Wende J, Stanford JB, Schisterman EF. Preconception Low-Dose Aspirin Restores Diminished Pregnancy and Live Birth Rates in Women With Low-Grade Inflammation: A Secondary Analysis of a Randomized Trial. J Clin Endocrinol Metab. 2017 May 1;102(5):1495-1504. doi: 10.1210/jc.2016-2917. PMID 28323989
- [Derived] Radin RG, Sjaarda LA, Perkins NJ, Silver RM, Chen Z, Lesher LL, Galai N, Wactawski-Wende J, Mumford SL, Schisterman EF. Low-Dose Aspirin and Sporadic Anovulation in the EAGeR Randomized Trial. J Clin Endocrinol Metab. 2017 Jan 1;102(1):86-92. doi: 10.1210/jc.2016-2095. PMID 27754808
- [Derived] Hinkle SN, Mumford SL, Grantz KL, Silver RM, Mitchell EM, Sjaarda LA, Radin RG, Perkins NJ, Galai N, Schisterman EF. Association of Nausea and Vomiting During Pregnancy With Pregnancy Loss: A Secondary Analysis of a Randomized Clinical Trial. JAMA Intern Med. 2016 Nov 1;176(11):1621-1627. doi: 10.1001/jamainternmed.2016.5641. PMID 27669539
- [Derived] Zarek SM, Mitchell EM, Sjaarda LA, Mumford SL, Silver RM, Stanford JB, Galai N, Schliep KC, Radin RG, Plowden TC, DeCherney AH, Schisterman EF. Antimullerian hormone and pregnancy loss from the Effects of Aspirin in Gestation and Reproduction trial. Fertil Steril. 2016 Apr;105(4):946-952.e2. doi: 10.1016/j.fertnstert.2015.12.003. Epub 2015 Dec 17. PMID 26707905
- [Derived] Zarek SM, Mitchell EM, Sjaarda LA, Mumford SL, Silver RM, Stanford JB, Galai N, White MV, Schliep KC, DeCherney AH, Schisterman EF. Is Anti-Mullerian Hormone Associated With Fecundability? Findings From the EAGeR Trial. J Clin Endocrinol Metab. 2015 Nov;100(11):4215-21. doi: 10.1210/jc.2015-2474. Epub 2015 Sep 25. PMID 26406293
- [Derived] Radin RG, Mumford SL, Silver RM, Lesher LL, Galai N, Faraggi D, Wactawski-Wende J, Townsend JM, Lynch AM, Simhan HN, Sjaarda LA, Perkins NJ, Zarek SM, Schliep KC, Schisterman EF. Sex ratio following preconception low-dose aspirin in women with prior pregnancy loss. J Clin Invest. 2015 Sep;125(9):3619-26. doi: 10.1172/JCI82357. Epub 2015 Aug 17. PMID 26280577
- [Derived] Silver RM, Ahrens K, Wong LF, Perkins NJ, Galai N, Lesher LL, Faraggi D, Wactawski-Wende J, Townsend JM, Lynch AM, Mumford SL, Sjaarda L, Schisterman EF. Low-dose aspirin and preterm birth: a randomized controlled trial. Obstet Gynecol. 2015 Apr;125(4):876-884. doi: 10.1097/AOG.0000000000000736. PMID 25751215
- [Derived] Schisterman EF, Mumford SL, Schliep KC, Sjaarda LA, Stanford JB, Lesher LL, Wactawski-Wende J, Lynch AM, Townsend JM, Perkins NJ, Zarek SM, Tsai MY, Chen Z, Faraggi D, Galai N, Silver RM. Preconception low dose aspirin and time to pregnancy: findings from the effects of aspirin in gestation and reproduction randomized trial. J Clin Endocrinol Metab. 2015 May;100(5):1785-91. doi: 10.1210/jc.2014-4179. Epub 2015 Feb 24. PMID 25710565
- [Derived] Schisterman EF, Silver RM, Lesher LL, Faraggi D, Wactawski-Wende J, Townsend JM, Lynch AM, Perkins NJ, Mumford SL, Galai N. Preconception low-dose aspirin and pregnancy outcomes: results from the EAGeR randomised trial. Lancet. 2014 Jul 5;384(9937):29-36. doi: 10.1016/S0140-6736(14)60157-4. Epub 2014 Apr 2. PMID 24702835
- See also: EAGeR Trial Home Page — https://www.nichd.nih.gov/about/org/diphr/eb/research/pages/effects-aspirin.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited using community-based advertisements and physician referral to four university medical centres in the US (2006-12).
Pre-assignment Details: Out of the 1397 women with confirmed eligibility, consented, and expressed initial interest in the study, 60 (4.3%) chose to discontinue the enrolment process. An additional 109 (7.8%) tested positive for pregnancy at the baseline visit or became pregnant before their randomisation visit.
Period: Overall Study
Arm/Group | Aspirin | Placebo
Started | 615 | 613
Completed | 535 | 543
Not Completed | 80 | 70
Not completed — Lost to Follow-up | 80 | 70

BASELINE CHARACTERISTICS:
Population: All women who consented and underwent randomization were included in baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | Placebo | Total
Number analyzed (Participants) | 615 | 613 | 1228
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (4.9) | 28.7 (4.7) | 28.7 (4.8)
Gender [Count of Participants; unit: Participants]
  Female | 615 | 613 | 1228
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 576 | 586 | 1162
  Non-White | 39 | 27 | 66

OUTCOME MEASURES:

1. Primary Outcome: Live Birth
Description: Live birth was obtained prospectively by maternal report and abstraction from medical records by trained staff .
Time Frame: after delivery
Population: Analyses were based on the intention-to-treat principle (excluding participants lost to follow-up).
Measure: Number; unit: livebirths
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 535 | 543
livebirths | 309 | 286
Statistical Analysis 1: Comparison: Aspirin vs Placebo; The study was designed to detect a 10% absolute difference in livebirth rate with 80% power and a type I error rate of 5%, on the assumption that participants taking placebo who achieved pregnancy would have a livebirth rate of 75%; Test type: Superiority or Other; p = 0.0984, Fisher Exact — Only one outcome for primary outcome, so no adjustment of p-value for multiple comparisons was done. A priori threshold for statistical significance was p<0.05; No adjustments were done. Treatment groups were similar with respect to the assessed demographic and baseline characteristics; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.98 to 1.22]

2. Secondary Outcome: hCG Recognized Pregnancy
Time Frame: within 8-weeks of gestation
Measure: Number; unit: pregnancy
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 535 | 543
pregnancy | 394 | 363
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = .0165, Fisher Exact; Risk Ratio (RR) = 1.10, 95% CI 2-sided [1.02 to 1.19]

3. Secondary Outcome: Clinically Recognized Pregnancy
Time Frame: 8-weeks
Measure: Number; unit: pregnancy
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 535 | 543
pregnancy | 374 | 346
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = .0329, Fisher Exact; Risk Ratio (RR) = 1.10, 95% CI 2-sided [1.01 to 1.19]

4. Secondary Outcome: Early Pregnancy Loss (EPL)
Description: Implantation failures
Time Frame: 8 weeks
Measure: Number; unit: pregnancy
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 537 | 551
pregnancy | 28 | 27
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = .8902, Fisher Exact; Risk Ratio (RR) = 1.06, 95% CI 2-sided [.64 to 1.78]

5. Secondary Outcome: Pregnancy Losses Occurring Less Than 10 Weeks
Description: Includes preembryonic and embryonic losses (exclusive of implantation failures)
Time Frame: less than 10-weeks
Measure: Number; unit: pregnancy
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 537 | 551
pregnancy | 56 | 53
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = .6869, Fisher Exact; Risk Ratio (RR) = 1.08, 95% CI 2-sided [.76 to 1.55]

6. Secondary Outcome: Fetal Pregnancy Loss
Time Frame: until 40 weeks
Measure: Number; unit: pregnancy
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 537 | 551
pregnancy | 4 | 6
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = .7530, Fisher Exact; Risk Ratio (RR) = .68, 95% CI 2-sided [.19 to 2.41]

7. Secondary Outcome: Stillbirth
Time Frame: 40 weeks
Measure: Number; unit: participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 537 | 551
participants | 2 | 2
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact; Risk Ratio (RR) = 1.03, 95% CI 2-sided [.15 to 7.26]

8. Secondary Outcome: Ectopic Pregnancy
Time Frame: within 6 weeks
Measure: Number; unit: pregnancy
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 537 | 551
pregnancy | 3 | 3
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact; Risk Ratio (RR) = 1.03, 95% CI 2-sided [.21 to 5.06]

9. Secondary Outcome: Molar Pregnancy
Time Frame: 8 weeks
Measure: Number; unit: pregnancy
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 535 | 543
pregnancy | 0 | 0
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact; Risk Ratio (RR) = 1.03, 95% CI 2-sided [.21 to 5.06]

10. Secondary Outcome: Preeclampsia
Time Frame: until delivery
Measure: Number; unit: participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 535 | 543
participants | 32 | 30
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = .7943, Fisher Exact; Risk Ratio (RR) = 1.08, 95% CI 2-sided [.67 to 1.76]

11. Secondary Outcome: Small for Gestational Age Infant
Description: birthweight
Time Frame: until delivery
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 535 | 543
grams | 3327 (521) | 3315 (550)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = .7802, t-test, 2 sided

12. Secondary Outcome: Preterm Birth
Time Frame: until delivery
Measure: Number; unit: infants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 535 | 543
infants | 22 | 31
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = .2603, Fisher Exact; Risk Ratio (RR) = .72, 95% CI 2-sided [.42 to 1.23]

13. Secondary Outcome: Abnormal Fetal Testing
Time Frame: 8 weeks
Population: No data were collected for this Outcome Measure.
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Fetal Intolerance of Labor
Time Frame: until delivery
Population: No data were collected for this Outcome Measure.
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Abruption
Description: Partial or complete abruption (ie, premature separation of the placenta)
Time Frame: until delivery
Measure: Number; unit: participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 615 | 613
participants | 7 | 5
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = 0.77, Fisher Exact; Risk Difference (RD) = 0.30, 95% CI 2-sided [-0.8 to 1.4]

ADVERSE EVENTS:
Arm/Group | Aspirin | Placebo
Serious Adverse Events (participants affected / at risk) | 7/615 | 5/613
Other Adverse Events (participants affected / at risk) | 24/615 | 8/613
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=615) | Placebo (N=613)
Transient Pulmonary Hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Minor Birth Defects (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 4 (4) — No difference was seen in the proportion of minor birth defects between the groups (four in each group). Of the four birth defects in the low dose aspirin group, one was a cleft lip and three were ventricular septal defects.
Neonatal Death (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) — Three cases of neonatal death occurred; of the two deaths in the lowdose aspirin group, one was due to cervical insufficiency and the other was attributed to chronic vaginal bleeding, chorioamnionitis, and preterm birth.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin (N=615) | Placebo (N=613)
Vaginal Bleeding (Pregnancy, puerperium and perinatal conditions) | 24 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes